CLINICAL TRIAL: NCT01792414
Title: Transcranial Electrical Stimulation (TES) for the Treatment of Depression.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HC12143
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active TES (Active Comparator): Active TES
  Interventions: Device: Active TES
- Sham TES (Sham Comparator): Sham TES
  Interventions: Device: Sham TES

INTERVENTIONS:
Device: Sham TES — Neuroconn Eldith device
  Arms: Sham TES
Device: Active TES — Neuroconn Eldith device
  Arms: Active TES

SUMMARY:
This study is a RCT of transcranial electrical stimulation in depressed patients. Mood, cognitive test performance and biomarkers will be measured during the trial.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depressive Episode (as part of a Major Depressive Disorder or Bipolar Disorder), of minimum 4 weeks duration.
* MADRS score ≥ 20 at study entry.

Exclusion Criteria:

* DSM-IV psychotic disorder;
* drug or alcohol abuse or dependence (preceding 12 months);
* inadequate response to ECT (current episode of depression);
* anticonvulsant or benzodiazepine medication;
* rapid clinical response required, e.g. high suicide risk; clinically defined neurological disorder or insult;
* metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites;
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 12 weeks

SECONDARY OUTCOMES:
Beck Depression Inventory II | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Black Dog Institute / University of New South Wales, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Nikolin S, Alonzo A, Martin D, Galvez V, Buten S, Taylor R, Goldstein J, Oxley C, Hadzi-Pavlovic D, Loo CK. Transcranial Random Noise Stimulation for the Acute Treatment of Depression: A Randomized Controlled Trial. Int J Neuropsychopharmacol. 2020 Apr 21;23(3):146-156. doi: 10.1093/ijnp/pyz072. PMID 31899509